CLINICAL TRIAL: NCT02622490
Title: Diet-induced Thermogenesis 2
Brief Title: Acute Effects of Different Macronutrient Compositions and Meal Distributions of the Food
Acronym: DIT2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Fredrik H Nystrom, professor, MD, University Hospital, Linkoeping
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DIT2
Record Dates: First submitted 2015-11-30; First posted 2015-12-04 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Metabolic Rate; Plasma Glucose; Serum Insulin; Serum Triglycerides; Sense of Satiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low carb. one meal (Active Comparator): Intervention: One meal of 750 kcal with 20 % of energy content from carbohydrates
  Interventions: Other: two test meals with two different macronutrient compositions
- Low Carb. 5 small meals (Active Comparator): Intervention: Five meals every 30 minutes of 150 kcal/each with 20 % of energy content from carbohydrates.
  Interventions: Other: two test meals with two different macronutrient compositions
- High carb. one meal (Active Comparator): Intervention: One meal of 750 kcal with 50 % of energy content from carbohydrates
  Interventions: Other: two test meals with two different macronutrient compositions
- High carb. 5 meals (Experimental): Intervention: Five meals every 30 minutes of 150 kcal/each with 50 % of energy content from carbohydrates.
  Interventions: Other: two test meals with two different macronutrient compositions

INTERVENTIONS:
Other: two test meals with two different macronutrient compositions — Either a high or a low carb meal either as one large or as 5 small meals. ie a crossover trial with one arm

SUMMARY:
About thirty participants, of varying degrees of obesity or being non-obese, without serious concomitant diseases consume either a high- or a low- carbohydrate beverage. The beverage is also consumed either as one single drink or as 5 small portions in the morning and are tested for effects on major cardiovascular risk markers and on metabolic rate for three hours on each occasion.

DETAILED DESCRIPTION:
Thirty participants come to the metabolic ward at about 8 o´clock in the fasting state and stay until lunch on four occasions each. The participants are randomized to the order of the test meals. The meals have a total caloric content of 750 kcal and have either 50% of energy from carbohydrates (low fat) or 20% of energy from carbohydrates (low carb.). The meals are consumed on one occasion in the morning or divided in 5 portions (150 kcal each) for every 30 minutes, i.e. total combinations of meal composition and of meal distribution is 4. Effects of the food on p-glucose, s-insulin, blood-lipids, hormones and on metabolic rate is measured by blood tests or by indirect calorimetry (for metabolic rate). Sense of satiety is measured by visual analogue scales.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants > 18 years with or without obesity

Exclusion Criteria:

* Major illnesses,
* thyroid diseases,
* need to take prednisolone,
* psychiatric disease,
* inability to understand Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-09; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Metabolic rate | During about 3 hours
  The metabolic rate is measured before (baseline) and there after repeatedly during 3 hours

SECONDARY OUTCOMES:
Effects on glucose and insulin | 3 hours
  Repeated test of glucose and insulin for three hours after test meal

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik H Nystrom, MD professor, Principal Investigator — Faculty of Medicine and Health Science, Linköping University, Sweden
Locations (1):
- University Hospital of Linkoping, Linköping, Sweden